CLINICAL TRIAL: NCT05392998
Title: Tolerance to Residual Astigmatism and Defocus in Eyes With a Non-diffractive Extended Depth of Focus (EDoF) Intraocular Lens
Brief Title: Tolerance to Residual Astigmatism in Eyes With Vivity®
Status: Completed | Type: Observational
Sponsor: Clínica Rementería (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 21/365-O_P_Viv
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Lenses, Intraocular
Keywords: extended depth of focus intraocular lens; astigmatism
MeSH Terms: conditions — Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Vivity patients: The study will include patients >40 years old that undergo routine cataract surgery and implantation of Vivity ®. Exclusion criteria include corneal astigmatism ≥1.0 diopters (D ), amblyopia, previous ocular surgery and presence of ocular pathologies and abnormal iris. Patients with intra- or postoperative complications, with a postoperative best distance corrected visual acuity (BDCVA) < 20/20 and with postoperative refractive astigmatism > 0.50D will be also excluded .
  Inclusion and exclusion criteria will be assessed by an ophthalmologic examination including refraction, screening for ocular conditions and/or systemic diseases, slit-lamp biomicroscopy and fundus examination.
  Interventions: Device: Cataract surgery with Vivity intraocular lens implantation

INTERVENTIONS:
Device: Cataract surgery with Vivity intraocular lens implantation — Cataract surgery with Vivity intraocular lens implantation

SUMMARY:
Low amounts of postoperative residual astigmatism may worsen the visual performance of patients implanted with presbyopia- correcting intraocular lenses (IOLs). Although extended depth of focus (EDoF) IOLS have introduced optical improvements, it is important to determine the tolerance of these IOLs to postoperative astigmatism. This is important for an appropriate surgical planning.

Therefore, the aim of this study is to simulate and assess the impact of mild amounts of residual mixed astigmatisms with the axis oriented in different positions (vertical, oblique and horizontal) in eyes implanted with the Vivity® IOL.

DETAILED DESCRIPTION:
Objectives:

* Primary objective: To describe the tolerance of simulated astigmatism on patients implanted with Vivity at far distance.
* Secondary objective: To describe the tolerance of simulated astigmatism on patients implanted with Vivity at intermediate distance.

Study Design: Prospective, single arm, descriptive, 3-month follow up.

Patient population: 30 consecutive eyes of 30 patients implanted with Vivity bilaterally with no postoperative complications. The calculation of the required sample size was based on monocular corrected distande visual acuity. A difference of 0.2 logMAR units was assumed to be clinically significant anda standard deviation of 0.05 was anticipated(data obtained from a comparative study between a bifocal and a trifocal IOL: Jonker SM, et al. Journal of Cataract Refract Surg. 2015; 41: 1631-40). Based on these assumptions, with an α of 0.05 and power of 0.8, it was calculated that 25 eyes were required in each group. Due to potential dropouts, a larger sample size has been selected.

Clinical Protocol: All patients fullfilling study criteria will be considered for inclusion three months after surgery. After patient consent, uncorrected distance visual acuity will be measured with an ETDRS chart, followed by subjective refraction (best distance correction). In all cases, mixed astigmatism will be induced with trial lens over the best distance corrected situation (considered the reference situation).

Once the best distance correction is determined, the different visual acuity evaluation procedures for this study will be performed with a Freiburg Acuity Test software package. The software will be run on a separate laptop screen calibrated to be presented at 4 meters. In this procedure, a black Landolt C is presented to the subjects and, among 8 different possibilities, they indicate the orientation of the optotype on a numeric keypad. This test minimizes the observer's bias because the presented optotype depends on the patient´s previous responses. That is, when the observer responds to a certain optotype, the software automatically modifies the size of the next optotype according to parameter estimation by a sequential test method. (7,8) Finally, all serious adverse events will be reported.

Statistical Analysis: Visual acuity values will be expressed as mean and standard deviation. Normal distribution of variables will be assessed using the Kolmogorov- Smirnov test. Pre- and post-operative data of each parameter will be compared by means of the Student's t-test. A repeated measure analysis of variance (ANOVA) will be used to gauge any statistically significant difference of the data within the different simulated situations. Differences are considered to be statistically significant for P value <0.05 (i.e., at the 5% level).

ELIGIBILITY:
Inclusion Criteria:

* Patients >40 years old that undergo routine cataract surgery
* Bilateral implantation of Vivity ® IOL

Exclusion Criteria:

* Corneal astigmatism ≥1.0 diopters (D )
* Amblyopia
* Previous ocular surgery
* Presence of ocular pathologies
* Abnormal iris
* Patients with intra- or postoperative complications
* Postoperative best distance corrected visual acuity (BDCVA) < 20/20
* Postoperative refractive astigmatism > 0.50D

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing bilateral cataract surgery with bilateral Vivity intraocular lens implantation, with no other ocular diseases and no complications
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laureano Rementeria-Capelo, MD, Principal Investigator — Clínica Rementería
Locations (1):
- Clínica Rementería, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after reasonable request

RESULTS

PARTICIPANT FLOW:
Groups:
- Vivity Patients: The study included patients >40 years old that underwent routine cataract surgery and IOL implantation. Exclusion criteria included corneal astigmatism ≥1.0 diopters (D), amblyopia, previous ocular surgery, and presence of ocular pathologies and abnormal iris. Patients with intra- or postoperative complications, with a postoperative distance corrected visual acuity (DCVA) <20/20 and with postoperative refractive astigmatism >0.50 D were also excluded.
Period: Overall Study
Arm/Group | Vivity Patients
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vivity Patients
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.37 (7.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Distance Against the Rule Astimatism
Description: Change from baseline condition in the monocular best corrected distance visual acuity, inducing astigmatism of +0.25-0.50x0*, taking as a reference the subjects' axis
Time Frame: Three months after surgery
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Vivity Patients
Number analyzed (Participants) | 30
LogMAR | 0.01 (0.04)

2. Primary Outcome: Distance Oblique Astigmatism
Description: Change from baseline condition in the monocular best corrected distance visual acuity, inducing astigmatism of +0.25-0.50x45*, taking as a reference the subjects' axis
Time Frame: Three months after surgery
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- Vivity Patients: The study will include patients >40 years old that undergo routine cataract surgery and implantation of Vivity ®. Exclusion criteria include corneal astigmatism ≥1.0 diopters (D ), amblyopia, previous ocular surgery and presence of ocular pathologies and abnormal iris. Patients with intra- or postoperative complications, with a postoperative best distance corrected visual acuity (BDCVA) < 20/20 and with postoperative refractive astigmatism > 0.50D will be also excluded .
  Inclusion and exclusion criteria will be assessed by an ophthalmologic examination including refraction, screening for ocular conditions and/or systemic diseases, slit-lamp biomicroscopy and fundus examination.
  Cataract surgery with Vivity intraocular lens implantation: Cataract surgery with Vivity intraocular lens implantation
Arm/Group | Vivity Patients
Number analyzed (Participants) | 30
LogMAR | 0.01 (0.06)

3. Primary Outcome: Distance With the Rule Astigmatism
Description: Change from baseline condition in the monocular best corrected distance visual acuity, inducing astigmatism of +0.25-0.50x90*, taking as a reference the subjects' axis
Time Frame: Three months after surgery
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Vivity Patients
Number analyzed (Participants) | 30
LogMAR | 0.01 (0.05)

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | Vivity Patients
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT05392998/Prot_SAP_000.pdf